CLINICAL TRIAL: NCT03162354
Title: Implementation Trial of a Validated Clinical Decision Rule for Pediatric Abusive Head Trauma (NIH Grant Number P50HD089922)
Brief Title: The CDR Implementation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kent Hymel, Child Abuse Pediatrician, Professor of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00005613; P50HD089922 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-22 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Pediatric Abusive Head Trauma

STUDY DESIGN:
Intervention Model Description: The stratified cluster randomized trial design will facilitate direct comparison of child abuse evaluations at four, randomly selected, control sites to four matched intervention sites, where investigators will deploy active, multifaceted, implementation strategies designed to promote CDR acceptability and application.
Who Masked: Outcomes Assessor
Masking Description: The study statistician will remain blinded to PICU site group membership (control vs. intervention sites).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Sites (Experimental): At the four intervention sites, investigators will deploy active, multifaceted, implementation strategies designed to promote CDR acceptability and application as an AHT screening tool. These strategies will include physician training with onsite visits, monthly "booster training emails," access to an "AHT probability calculator," audit and site-specific feedback, and local "information sharing sessions" designed to address local barriers to CDR acceptance and application.
  Interventions: Other: Application of a validated Clinical Decision Rule (CDR) as an AHT screening tool
- Control Sites (No Intervention): At the four matched control sites, physicians will engage in "AHT screening as usual."

INTERVENTIONS:
Other: Application of a validated Clinical Decision Rule (CDR) as an AHT screening tool — The Clinical Decision Rule (CDR) for AHT reads as follows:
  Every acutely head-injured infant or young child hospitalized for intensive care presenting with any one or more of these four variables should be considered "high risk" and thoroughly evaluated for abuse: (1) any clinically significant respiratory compromise at the scene of injury, during transport, in the Emergency Department, or prior to admission; (2) Any bruising involving the child's ear(s), neck, or torso; (3) Any subdural hemorrhage(s) or fluid collection(s) that are bilateral OR involve the interhemispheric space; (4) Any skull fracture(s) other than an isolated, nondiastatic, linear, parietal, skull fracture.
  Arms: Intervention Sites

SUMMARY:
To increase the accuracy of doctors' decisions to launch or forgo child abuse evaluations in their young, acutely head-injured patients, investigators have derived and validated a clinical decision rule (CDR) that detects abusive head trauma (AHT) with 96% sensitivity in pediatric intensive care unit (PICU) settings. This "CDR Implementation Trial" across eight PICU sites will assess the CDR's actual impact on AHT screening accuracy, identify factors associated with maximal physician acceptance and application of this novel AHT screening tool, and assess the sustainability of active CDR implementation strategies.

DETAILED DESCRIPTION:
Investigators' long-term goal is to increase the accuracy of doctors' decisions to launch or forgo child abuse evaluations in their young, acutely head-injured patients. To this end, PediBIRN investigators have derived and validated a 4-variable clinical decision rule (CDR) that detects abusive head trauma (AHT) with 96% sensitivity in PICU settings. Applied at PICU admission, the CDR categorizes young, acutely head-injured patients as higher risk vs. lower risk, and recommends thorough abuse evaluations for all higher risk patients.

The "CDR Implementation Trial" across eight PICUs will assess the CDR's actual impact on AHT screening accuracy. The stratified cluster randomized trial design will facilitate direct comparison of child abuse evaluations at four, randomly selected, control sites to four matched intervention sites, where investigators will deploy active, multifaceted, implementation strategies designed to promote CDR acceptability and application. These strategies will include physician training with onsite visits, monthly "booster training emails," access to an "AHT probability calculator," audit and site-specific feedback, and local "information sharing sessions" designed to address local barriers to CDR acceptance and application.

PediBIRN investigators will conduct the CDR Implementation Trial with three Specific Aims. Aim 1 is to assess the CDR's actual impact on AHT screening accuracy. Investigators hypothesize that deployment of CDR implementation strategies at the four intervention sites will be associated with higher percentages of higher risk patients evaluated thoroughly for abuse, and lower percentages of lower risk patients evaluated (even partially) for abuse. Aim 2 is to identify factors that impact CDR application in PICU settings. Investigators hypothesize that PICUs with higher patient volumes, providers with child abuse expertise, and providers with more intense exposure to CDR implementation strategies will be predictive of higher percentages of higher risk patients thoroughly evaluated for abuse, whereas patients of minority race or ethnicity will be predictive of higher percentages of lower risk patients evaluated for abuse. Investigators' third Exploratory Aim is to measure the sustained impacts of CDR implementation strategies. Investigators hypothesize that CDR utilization at intervention sites will be sustained twelve months after CDR implementation strategies have been discontinued.

Based on strong Preliminary Studies, investigators predict that CDR adoption as an AHT screening tool will increase AHT detection; reduce overall abuse evaluations and their associated risks; reduce unwarranted variation in current AHT screening practices; minimize the adverse impacts of doctors' inherent biases, uncertainty, and practice disparities; reduce AHT-associated acute health care costs in PICU settings; and save the lives of children who will be reinjured and killed if their AHT is missed or unrecognized.

ELIGIBILITY:
Inclusion Criteria:

* Children under 3 years of age admitted to a PICU for management of symptomatic, acute, closed, traumatic, cranial, or intracranial injuries confirmed by computed tomography (CT) or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Patients admitted to a PICU with acute head injuries resulting from a collision involving a motor vehicle.
* Patients admitted to a PICU with acute head injuries and clear evidence on neuroimaging of pre-existing brain malformation, disease, infection, or hypoxia-ischemia.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent P. Hymel, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (8):
- United States (8):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Wesley Hospital, Wichita, Kansas
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Cneter and Children's Hospital of Omaha, Omaha, Nebraska
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - University of Texas health Sciences Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Richmond, Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hymel KP, Willson DF, Boos SC, Pullin DA, Homa K, Lorenz DJ, Herman BE, Graf JM, Isaac R, Armijo-Garcia V, Narang SK; Pediatric Brain Injury Research Network (PediBIRN) Investigators. Derivation of a clinical prediction rule for pediatric abusive head trauma. Pediatr Crit Care Med. 2013 Feb;14(2):210-20. doi: 10.1097/PCC.0b013e3182712b09. PMID 23314183
- [Background] Hymel KP, Armijo-Garcia V, Foster R, Frazier TN, Stoiko M, Christie LM, Harper NS, Weeks K, Carroll CL, Hyden P, Sirotnak A, Truemper E, Ornstein AE, Wang M; Pediatric Brain Injury Research Network (PediBIRN) Investigators. Validation of a clinical prediction rule for pediatric abusive head trauma. Pediatrics. 2014 Dec;134(6):e1537-44. doi: 10.1542/peds.2014-1329. Epub 2014 Nov 17. PMID 25404722
- [Background] Hymel KP, Herman BE, Narang SK, Graf JM, Frazier TN, Stoiko M, Christie LM, Harper NS, Carroll CL, Boos SC, Dias M, Pullin DA, Wang M; Pediatric Brain Injury Research Network (PediBIRN) Investigators; Pediatric Brain Injury Research Network PediBIRN Investigators. Potential Impact of a Validated Screening Tool for Pediatric Abusive Head Trauma. J Pediatr. 2015 Dec;167(6):1375-81.e1. doi: 10.1016/j.jpeds.2015.09.018. Epub 2015 Oct 23. PMID 26477871
- [Derived] Hymel KP, Armijo-Garcia V, Musick M, Marinello M, Herman BE, Weeks K, Haney SB, Frazier TN, Carroll CL, Kissoon NN, Isaac R, Foster R, Campbell KA, Tieves KS, Livingston N, Bucher A, Woosley MC, Escamilla-Padilla D, Jaimon N, Kustka L, Wang M, Chinchilli VM, Dias MS, Noll J; Pediatric Brain Injury Research Network (PediBIRN) Investigators. A Cluster Randomized Trial to Reduce Missed Abusive Head Trauma in Pediatric Intensive Care Settings. J Pediatr. 2021 Sep;236:260-268.e3. doi: 10.1016/j.jpeds.2021.03.055. Epub 2021 Mar 31. PMID 33798512
- See also: Website for "The CDR Implementation Trial" — http://www.pedibirn.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participating PICUs were stratified based on projected patient volumes, matched into pairs, and allocated randomly to intervention (n=4) or control (n=4) conditions. Eligible participants were acutely head injured patients <3 years admitted for intensive care (excluding MVA victims and patients with pre-existing brain abnormalities). Prospective data capture at all 8 participating PICUs began 1 August 2017 and ended 31 March 2020. For patients, the study was strictly observational.
Pre-assignment Details: All eligible patients were included in the analysis.
Units Other Than Participants: Pediatric intensive care units
Groups:
- Intervention Sites: At the four intervention sites, investigators will deploy active, multifaceted, implementation strategies designed to promote CDR acceptability and application as an AHT screening tool. These strategies will include physician training with onsite visits, monthly "booster training emails," access to an "AHT probability calculator," audit and site-specific feedback, and local "information sharing sessions" designed to address local barriers to CDR acceptance and application.
  Application of a validated Clinical Decision Rule (CDR) as an AHT screening tool: The Clinical Decision Rule (CDR) for AHT reads as follows:
  Every acutely head-injured infant or young child hospitalized for intensive care presenting with any one or more of these four variables should be considered "high risk" and thoroughly evaluated for abuse: (1) any clinically significant respiratory compromise at the scene of injury, during transport, in the Emergency Department, or prior to admission; (2) Any bruising involving the child's ear(s), neck, or torso; (3) Any subdural hemorrhage(s) or fluid collection(s) that are bilateral OR involve the interhemispheric space; (4) Any skull fracture(s) other than an isolated, nondiastatic, linear, parietal, skull fracture.
Period: Overall Study
Arm/Group | Intervention Sites | Control Sites
Started | 183; 4 Pediatric intensive care units | 237; 4 Pediatric intensive care units
Completed | 183; 4 Pediatric intensive care units | 237; 4 Pediatric intensive care units
Not Completed | 0; 0 Pediatric intensive care units | 0; 0 Pediatric intensive care units

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Sites | Control Sites | Total
Number analyzed (Participants) | 183 | 237 | 420
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.7 (7.2) | 8.7 (8.8) | 8.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 87 | 155
  Male | 115 | 150 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 88 | 109
  Not Hispanic or Latino | 142 | 127 | 269
  Unknown or Not Reported | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 43 | 37 | 80
  White | 99 | 174 | 273
  More than one race | 12 | 7 | 19
  Unknown or Not Reported | 25 | 14 | 39
Region of Enrollment [Number; unit: participants]
  United States | 183 | 237 | 420
Higher Risk [Number; unit: participants] — To reduce cases of missed or unrecognized abusive head trauma (AHT), Pediatric Brain Injury Research Network (PediBIRN) investigators derived and validated an AHT screening tool. The screening tool comes in the form of a directive, 4-variable, clinical decision rule (CDR). The "PediBIRN-4" CDR stratifies patients as "higher risk" vs. "lower risk" and recommends that every higher risk patient be thoroughly evaluated for abuse. Higher risk patients were those who presented for intensive care with any one or more of the CDR's four predictor variables.
  participants | 158 | 175 | 333
Lower Risk [Number; unit: participants] — To reduce cases of missed or unrecognized abusive head trauma (AHT), Pediatric Brain Injury Research Network (PediBIRN) investigators derived and validated an AHT screening tool. The screening tool comes in the form of a directive, 4-variable, clinical decision rule (CDR). The "PediBIRN-4" CDR stratifies patients as "higher risk" vs. "lower risk." Lower risk patients were those who presented for intensive care with none of the CDR's four predictor variables. The CDR makes no recommendations regarding abuse evaluations of the patients it stratifies as lower risk.
  participants | 25 | 62 | 87

OUTCOME MEASURES:

1. Primary Outcome: The Number of Higher Risk Patients Evaluated Thoroughly for Abuse at Intervention vs. Control Sites
Description: This outcome measure facilitates a comparison of the percentage of patients that the clinical decision rule stratified as higher risk who were evaluated thoroughly for abuse (with both skeletal survey and retinal exam) at intervention vs. control sites. We hypothesized that thorough evaluations of higher risk patients would be significantly higher at intervention sites.
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From all patients in each arm of the trial that the clinical prediction rule specified to be at higher risk for abuse, this outcome measures the proportion that were evaluated "thoroughly" for abuse with skeletal survey AND retinal exam by an ophthalmologist.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 158 | 175
Participants | 128 | 128
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; We powered this hypothesis to detect a 17% increase (from 73% to 90%) in higher risk patients evaluated thoroughly for abuse at intervention sites, compared to baseline in prior PediBIRN studies. Generalized linear mixed-effects models were adopted to analyze 1,000 Monte Carlo datasets from simulation. For the target sample size of 304 higher risk patients (152 in each arm), the proportion of simulated datasets that yielded a statistically significant result for the primary hypothesis was 95.7%; Test type: Other; p = 0.11, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.37 to 1.11] — The direction of the comparison is from intervention sites to control sites

2. Primary Outcome: The Number of Lower Risk Patients Evaluated Even Partially for Abuse at Intervention vs. Control Sites
Description: This outcome measure facilitates a comparison of the percentage of patients that the clinical decision rule stratified as lower risk who were nevertheless evaluated at least partially for abuse (with skeletal survey and/or retinal examination) at intervention vs. control sites. We hypothesized that (partial or complete) abuse evaluations of lower risk patients would be significantly lower at intervention sites.
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From all patients in each arm of the trial that the clinical prediction rule specified to be at lower risk for abuse, this outcome measures the proportion that were (nevertheless) evaluated even partially for abuse with skeletal survey and/or retinal exam by an ophthalmologist.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 25 | 62
Participants | 17 | 37
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.49, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.24 to 1.98] — The direction of the comparison is from intervention sites to control sites

3. Primary Outcome: Estimated Rates (Percentages) of Missed AHT at Intervention vs. Control Sites
Description: This outcome measures and compares estimated rates (percentages) of missed AHT (among all patients with AHT) at intervention vs. control sites. Using secondary outcome measures, it was calculated as [estimated cases of missed AHT] / [estimated cases of missed AHT + patients with corroborating findings of abuse]. We hypothesized that the estimated rate of missed AHT would be significantly lower at intervention sites. This outcome measure is best interpreted in the following contexts: (1) Applied accurately and consistently, the clinical decision rule's potential sensitivity for AHT is 96% (see references). That is, it should "miss" (categorize as lower risk) only 4% of AHT patients, and (2) We estimate that intervention and control site physicians "missed" 15% and 11% of their AHT patients, respectively, in prior PediBIRN studies (see the Post-Hoc Outcome "The Estimated Rate of Missed AHT at Intervention vs. Control Sites in Prior PediBIRN Studies").
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From those patients deemed to be victims of AHT in each arm of the trial, this outcome estimates the proportion whose AHT may have been missed or unrecognized.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 81 | 107
Participants | 6 | 14
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.22, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.69 to 5.13] — The direction of the comparison is from intervention sites to control sites

4. Secondary Outcome: The Number of Patients Evaluated at Least Partially for Abuse at Intervention vs. Control Sites
Description: This outcome measure facilitates a comparison of the percentage of patients evaluated at least partially for abuse (with skeletal survey and/or retinal examination) at intervention vs. control sites. Thus, it facilitates a broad-based comparison of AHT evaluation practices at intervention vs. control sites.
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From all eligible patients in each arm of the trial, this outcome measures the proportion who were evaluated at least partially for abuse with skeletal survey and/or retinal examination by an ophthalmologist.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 183 | 237
Participants | 163 | 189
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.01, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.27 to 0.85] — The direction of the comparison is from intervention sites to control sites

5. Secondary Outcome: The Number of Patients With Corroborating Findings of Abuse at Intervention vs. Control Sites (Aka Overall Diagnostic Yield)
Description: This outcome measure facilitates a comparison of the percentage of patients whose completed skeletal surveys and/or retinal exams revealed findings considered moderately or highly specific for abuse at intervention vs. control sites. Thus, it is also a measure of the overall diagnostic yield of patients' completed skeletal surveys and retinal examinations.
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From all patients in each arm of the trial who underwent at least a partial evaluation for abuse, this outcome measures the proportion whose completed skeletal survey and/or retinal examination by an ophthalmologist revealed moderately or highly specific findings of abuse.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 163 | 189
Participants | 75 | 93
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.84, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.46 to 2.60] — The direction of the comparison is from intervention sites to control sites

6. Secondary Outcome: The Number of Potential Cases of Missed AHT at Intervention vs. Control Sites
Description: This outcome measure facilitates a comparison of the percentage of eligible patients who might be potential cases of missed AHT (that is, patients lacking skeletal survey and/or retinal exam, whose abuse evaluation is therefore incomplete) at intervention vs. control sites.
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From all eligible patients in each arm of the trial, this outcome measures the proportion of patients that are potential cases of missed AHT (i.e., patients not evaluated for abuse, and, patients with negative incomplete abuse evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 183 | 237
Participants | 38 | 75
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.05, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.00 to 3.38] — The direction of the comparison is from intervention sites to control sites

7. Secondary Outcome: The Number of Estimated Patients With Missed AHT at Intervention vs. Control Sites
Description: This outcome measure facilitates a comparison of the estimated percentage of patients with missed AHT (among potential cases of missed AHT) at intervention vs. control sites. It was calculated as [potential cases of missed AHT] x [their mean estimate of abuse probability]. The patient-specific estimates of abuse probability used to calculate the mean estimates were accessed by applying the 4-variable rule as a clinical prediction tool (rather than a directive decision rule).
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From patients in each arm of the trial who are potential cases of missed abuse, this outcome measures the proportion of patients whose AHT may have been missed or unrecognized.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 38 | 75
Participants | 6 | 14
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.71, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.43 to 3.49] — The direction of the comparison is from intervention sites to control sites

8. Secondary Outcome: Estimated Prevalence of AHT at Intervention vs. Control Sites
Description: This outcome measure facilitates a comparison of the estimated prevalence of AHT (among all eligible patients) at intervention vs. control sites. It was calculated as [patients with corroborating findings of abuse + estimated cases of missed AHT] / [all eligible patients in each arm of the trial].
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From all eligible patients in each arm of the trial, this outcome estimates the proportion who were victims of AHT.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 183 | 237
Participants | 81 | 107
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.86, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.70 to 1.53] — The direction of the comparison is from intervention sites to control sites

9. Other Pre Specified Outcome: The Change (From Prior PediBIRN Studies to the Current Clinical Trial) in the Number of Higher Risk Patients Evaluated Thoroughly for Abuse at Intervention Sites
Description: This outcome measure facilitates a comparison of the percentage of higher risk patients evaluated thoroughly for abuse (with skeletal survey AND retinal examination) at intervention sites in prior strictly observational PediBIRN studies vs. the current cluster randomized trial. It was calculated using precisely equivalent methods and data captured prospectively between 2010 and 2013 in comparable patient cohorts at the same four intervention sites.
Time Frame: To be measured 32 months after the start of the clinical trial
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Sites at Baseline: Equivalent, eligible, young, acutely head-injured patients hospitalized for intensive care at one of the same four intervention sites during prior PediBIRN studies, conducted between 2010 and 2013.
- Intervention Sites During the Cluster Randomized Trial: At the four intervention sites, investigators will deploy active, multifaceted, implementation strategies designed to promote CDR acceptability and application as an AHT screening tool. These strategies will include physician training with onsite visits, monthly "booster training emails," access to an "AHT probability calculator," audit and site-specific feedback, and local "information sharing sessions" designed to address local barriers to CDR acceptance and application.
Arm/Group | Intervention Sites at Baseline | Intervention Sites During the Cluster Randomized Trial
Number analyzed (Participants) | 132 | 158
Participants | 89 | 128
Statistical Analysis 1: Comparison: Intervention Sites at Baseline vs Intervention Sites During the Cluster Randomized Trial; Test type: Other; p = 0.01, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.16 to 3.52] — The direction of the comparison is from baseline prior studies to the cluster randomized trial

10. Other Pre Specified Outcome: The Change (From Prior PediBIRN Studies to the Current Clinical Trial) in the Number of Potential Cases of Missed AHT at Intervention Sites
Description: This outcome measure facilitates a comparison of the percentage of potential cases of missed AHT (among all eligible patients) at intervention sites in prior strictly observational PediBIRN studies vs. the current cluster randomized trial. It was calculated using precisely equivalent methods and data captured prospectively between 2010 and 2013 in comparable patient cohorts at the same four intervention sites.
Time Frame: To be measured 32 months after the start of the clinical trial
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites at Baseline | Intervention Sites During the Cluster Randomized Trial
Number analyzed (Participants) | 172 | 183
Participants | 68 | 38
Statistical Analysis 1: Comparison: Intervention Sites at Baseline vs Intervention Sites During the Cluster Randomized Trial; Test type: Other; p < .001, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.26 to 0.67] — The direction of the comparison is from baseline in prior studies to the cluster randomized trial

11. Other Pre Specified Outcome: The Change (From Prior PediBIRN Studies to the Current Clinical Trial) in the Estimated Rate (Percentage) of Missed AHT at Intervention Sites
Description: This outcome measure facilitates a comparison of the estimated rate (percentage) of missed AHT (among all patients with AHT) at intervention sites in prior strictly observational PediBIRN studies vs. the current cluster randomized trial. It was calculated using precisely equivalent methods and data captured prospectively between 2010 and 2013 in comparable patient cohorts at the same four intervention sites.
Time Frame: To be measured 32 months after the start of the clinical trial
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites at Baseline | Intervention Sites During the Cluster Randomized Trial
Number analyzed (Participants) | 74 | 81
Participants | 11 | 6
Statistical Analysis 1: Comparison: Intervention Sites at Baseline vs Intervention Sites During the Cluster Randomized Trial; Test type: Other; p = 0.14, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.16 to 1.31] — The direction of the comparison is from baseline in prior PediBIRN studies to the clinical trial

12. Other Pre Specified Outcome: The Number of AHT Patients (Among All Patients With AHT) That the CDR Would Have Stratified as Higher Risk if the CDR Had Been Applied Accurately and Consistently (Aka the Clinical Decision Rule's Potential AHT Screening Sensitivity)
Description: This outcome measure facilitates estimation of the clinical decision rule's potential AHT screening sensitivity IF it had been applied accurately and consistently across all eight participating sites. It was calculated based on the following assumptions: (1) All higher risk patients were evaluated thoroughly for abuse with skeletal survey AND retinal exam by an ophthalmologist; Therefore, all cases of AHT among higher risk patients were recognized, and (2) Abuse evaluations were deferred in all lower risk patients; Therefore, all cases of AHT among lower risk patients were missed or unrecognized.
Time Frame: To be measured 32 months after the start of the clinical trial
Measure: Count of Participants; unit: Participants
Groups:
- All Eight Participating Sites: The four intervention sites and four control sites
Arm/Group | All Eight Participating Sites
Number analyzed (Participants) | 188
Participants | 181

13. Post Hoc Outcome: The Estimated Rate (Percentage) of Missed AHT at Intervention vs. Control Sites in Prior PediBIRN Studies
Description: This outcome facilitates comparison of the estimated rates (percentages) of missed AHT (among all patients with AHT) at intervention vs. control sites in prior strictly observational PediBIRN studies. It was calculated using precisely equivalent methods and data captured in comparable patient cohorts at the same eight sites between 2010 and 2013. The results provide context for interpreting estimated rates of missed AHT during the subsequent cluster randomized trial.
Time Frame: To be measured 32 months after the start of the clinical trial.
Population: From those patients deemed to be victims of AHT, in prior PediBIRN studies, at the same PICU sites that are participating in each arm of the current trial, this outcome estimates the proportion whose AHT may have been missed or unrecognized.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Sites: At the same four intervention sites, during prior (strictly observational) PediBIRN studies conducted to derive and validate the PediBIRN 4-variable clinical decision rule.
- Control Sites: At the same four control sites, during prior (strictly observational) PediBIRN studies conducted to derive and validate the PediBIRN 4-variable clinical decision rule.
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 74 | 61
Participants | 11 | 7
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.57, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.27 to 2.05] — The direction of the comparison is from intervention sites to control sites

14. Post Hoc Outcome: The Number of Potential Cases of Missed AHT at Intervention vs. Control Sites in Prior PediBIRN Studies
Description: This outcome measure facilitates comparison of the percentage of potential cases of missed AHT (among all eligible patients) in prior strictly observational PediBIRN studies at intervention vs. control sites. It was calculated using precisely equivalent methods and data captured in comparable patient cohorts at the same eight sites between 2010 and 2013. The results provide context for interpreting estimated rates of missed AHT during the subsequent cluster randomized trial.
Time Frame: To be measured 32 months after the start of the clinical trial
Population: From all eligible patients hospitalized in prior PediBIRN studies at the same PICU sites participating in each arm of the current trial, this outcome measures the proportion who represent potential cases of missed AHT.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Sites | Control Sites
Number analyzed (Participants) | 172 | 165
Participants | 68 | 48
Statistical Analysis 1: Comparison: Intervention Sites vs Control Sites; Test type: Other; p = 0.04, Chi-squared — The threshold for statistical significance was p = 0.05; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.40 to 0.99] — The direction of the comparison is from intervention sites to control sites

ADVERSE EVENTS:
Time Frame: 32 months
Arm/Group | Intervention Sites | Control Sites
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/237
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/237
Other Adverse Events (participants affected / at risk) | 0/183 | 0/237

LIMITATIONS AND CAVEATS:
CDR implementation supports may not have been delivered uniformly. We relied on imperfect patient-specific estimates of AHT probability to predict the results of abuse evaluations never completed. We failed to capture prospective data that might explain absent or incomplete abuse evaluations (e.g., early death). The trial was likely underpowered. Our results are not generalizable to non-PICU settings, to PICUs in non-academic centers, or to PICUs lacking access to CAP physicians.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03162354/Prot_SAP_000.pdf